CLINICAL TRIAL: NCT01972516
Title: A Phase II Study of Tivozanib as Maintenance Therapy, Post-Chemotherapy, in Patients With Platinum-Sensitive Ovarian, Fallopian Tube, or Primary Peritoneal Cancer
Brief Title: Tivozanib As Maintenance Therapy In GYN
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: due to slow accrual
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: National Comprehensive Cancer Network (Network); AVEO Pharmaceuticals, Inc. (Industry)
Responsible Party: Principal Investigator, Susana M. Campos, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 13-375
Record Dates: First submitted 2013-10-24; First posted 2013-10-30 (Estimated); Results first posted 2016-08-24 (Estimated); Last update posted 2017-06-05 (Actual); Status verified 2017-05

CONDITIONS: Ovarian Cancer; Fallopian Tube Cancer; Primary Peritoneal Carcinoma
Keywords: Platinum-Sensitive; Ovarian Cancer; Fallopian Tube Cancer; Primary Peritoneal Cancer; High-grade Serous
MeSH Terms: conditions — Ovarian Neoplasms; Fallopian Tube Neoplasms | interventions — tivozanib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tivozanib (Experimental): Tivozanib hydrochloride will be administered orally, at a dose of 1.5 mg/day, beginning on Day 1 of Cycle 1. Subjects will receive tivozanib hydrochloride once daily for 3 weeks followed by 1 week off treatment. One cycle is defined as 4 weeks. Cycles will be repeated every 4 weeks in the absence of disease progression or unacceptable toxicities.
  Interventions: Drug: Tivozanib
- Standard Care (No Intervention): Participants in the non-interventional arm will not receive study treatment, and will receive standard clinical observation and study assessments. Patients will continue to be observed in the absence of disease progression or unacceptable toxicities.

INTERVENTIONS:
Drug: Tivozanib
  Other Names: Tivozanib hydrochloride; AV-951
  Arms: Tivozanib

SUMMARY:
This research study is evaluating a drug called tivozanib as a possible treatment for ovarian, fallopian tube or primary peritoneal cancer.

Angiogenesis is the formation of new blood vessels. Tumors need blood vessels to grow and spread. Tivozanib is an anti-angiogenesis medicine that fights cancer by cutting off a tumor's blood supply so that it does not get the blood and nutrients it needs to grow.

In this research study, the Investigators are looking to see whether tivozanib works as a maintenance therapy for ovarian, fallopian tube or primary peritoneal carcinoma in participants who have achieved a complete response following chemotherapy. Maintenance therapy is given after a disease has responded to previous treatment. It is given to help prevent the spread or recurrence of the tumor.

DETAILED DESCRIPTION:
Once the participant has signed the consent form, they will be asked to undergo some screening tests or procedures to find out if the participant can be in the research study. Many of these tests and procedures are likely to be part of regular cancer care and may be done even if it turns out that the participant do not take part in the research study. If the participant has had some of these tests or procedures recently, they may or may not have to be repeated.

* A medical history, which includes questions about the participant's health, current medications, and any allergies.
* Performance status, which evaluates how the participant is able to carry on with their usual activities.
* A tumor assessment by CT (Computerized Tomography) scan or MRI (Magnetic Resonance Imaging.
* Blood tests.
* Urine test.
* Electrocardiogram (ECG)

If these tests show that the participant is eligible to participate in the research study, the participant will begin the study treatment. If the participant does not meet the eligibility criteria, the participant will not be able to participate in this research study.

Additional research procedures to be performed during this study:

- Archival tumor testing: During this study, additional tests will be performed on a sample of the participant's original tumor that has been stored in the institution's tissue banks. These tests will be performed on tumor tissue samples from previous biopsies or surgeries for the participant's cancer.

The research done on these samples will involve looking at DNA and proteins in the participant's cancer to see if researchers can learn more about the participant's type of cancer and understand how tivozanib might work on their tumor. Testing of this sample will not require the participant to undergo any additional research procedures.

This research sample collection is a required part of this research study.

Tissue collection / Ownership: Participation in this protocol involves providing specimen(s) of participant's tissue. Please know that if the investigator leaves the institution, the research and the tissue might remain at the DF/HCC or might be transferred to another institution.

After the screening procedures confirm that the participant are eligible to participate in the research study:

If the participant takes part in this research study, the participant will be randomized to receive tivozanib by mouth or no therapy. The participant will be given a study drug diary for each treatment if the participant is randomized to the tivozanib group.

Each treatment cycle lasts 28 days (4 weeks). For participants who are randomized to receive tivozanib, the participant will be taking the study drug once per day for 3 weeks followed by a week of rest. The diary will also include special instructions for taking the study drug. The study drug will be taken once a day with plenty of water.

ELIGIBILITY:
Inclusion Criteria:

* No evidence of disease on CT/MRI following treatment for recurrent ovarian, fallopian tube, or peritoneal cancer.
* High-grade papillary serous carcinoma of the ovary, fallopian tube or peritoneum. Histological confirmation of the original primary tumor is required.
* CA-125 within normal range.
* Age greater than or equal to 18 years.
* 1 prior line of therapy (cytotoxic therapy only) in the recurrent setting is allowed. Bevacizumab in the upfront setting allowed, however Bevacizumab or other VEGF pathway targeted therapy in the recurrent setting is not allowed. Hormonal therapy does not count as a prior line.
* Recovered from effects of recent surgery, radiotherapy, and chemotherapy.
* ECOG performance status ≤ 2

Organ and marrow function as defined below:

* Absolute neutrophil count ≥1,250/mcL
* Platelets ≥100,000/mcL
* Bilirubin ≤ 1.5 x ULN
* AST (SGOT) / ALT (SGPT) ≤ 2.5 x institutional upper limit of normal Alkaline phosphatase ≤ to 2.5 x ULN
* Creatinine ≤ 1.5 x institutional upper limit
* Less than or equal to 1+ proteinuria on two consecutive dipsticks taken no less than 1 week apart, or < 1 gm protein on 24-hour urine collection or a urine protein:creatinine ratio of < 1.
* INR < 1.5; if on anticoagulation: INR is required to be between 2 and 3.

Patient must receive one of these three regimens for their platinum sensitive disease (number of cycles should not have exceeded 8 cycles of 1 regimen in the recurrent setting):

* Platinum (Carboplatin or Cisplatin) and Taxane (Paclitaxel or Docetaxel) Carboplatin and Gemcitabine
* Carboplatin and Liposomal Doxorubicin
* Females not of childbearing potential or has documentation of a negative pregnancy test prior to the start of the study treatment are eligible. Sexually active pre-menopausal female subjects must agree to use adequate, highly effective contraceptive measures, while on study and for 45 days after the last dose of last study drug. Effective birth control includes (a) intrauterine device (IUD) plus one barrier method; (b) oral, implantable or injectable contraceptives plus one barrier method; or (c) 2 barrier methods. Effective barrier methods are male or female condoms, diaphragms, and spermicides (creams or gels that contain a chemical to kill sperm).
* Able and willing to sign a written informed consent document.

Exclusion Criteria:

* Prior therapy with bevacizumab or other VEGF pathway targeted therapy in the recurrent setting. Bevacizumab in the upfront setting is allowed.
* Receiving any other study agents.
* Subjects with treated limited stage basal cell or squamous cell carcinoma of the skin or carcinoma in situ of the breast or cervix are eligible. Subjects with prior cancer treated with a curative intent with no evidence of recurrent disease 5 years following diagnosis and judged by the investigator to be at low risk of recurrence are eligible. Subjects with any other concomitant or prior malignancies are ineligible.
* Serious non-healing wounds or ulcers at the time of registration.
* History of abdominal fistula or gastrointestinal perforation.
* Active bleeding.
* Clinically significant cardiovascular disease.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to Tivozanib.
* Symptomatic left ventricular dysfunction or baseline left ventricular ejection fraction (LVEF) by multigated acquisition scan (MUGA) or echocardiogram (ECHO) ≤ 50 % lower limit of institutional normal (LLN).
* Uncontrolled hypertension: systolic blood pressure of >140 mmHg or diastolic blood pressure of >90 mmHg documented on 2 consecutive measurements taken at least 24 hours apart.
* Myocardial infarction, severe angina, or unstable angina within 6 months prior to administration of first dose of study drug.
* History of serious ventricular arrhythmia (i.e., ventricular tachycardia or ventricular fibrillation).
* Cardiac arrhythmias requiring anti-arrhythmic medications (except for atrial fibrillation that is well controlled with anti-arrhythmic medication).
* Coronary or peripheral artery bypass graft within 6 months of screening.
* History of Class III or IV congestive heart failure, as defined by the New York Heart Association.
* Central nervous system metastases.

Note: Subjects with previously treated (radiotherapy or surgery) brain metastasis that have been stable without steroid treatment for at least 3 months following prior treatment may be enrolled.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2013-11; Primary Completion 2015-07 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susana Campos, MD, MPH, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana-Farber Cancer Institute, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Gaitskell K, Rogozinska E, Platt S, Chen Y, Abd El Aziz M, Tattersall A, Morrison J. Angiogenesis inhibitors for the treatment of epithelial ovarian cancer. Cochrane Database Syst Rev. 2023 Apr 18;4(4):CD007930. doi: 10.1002/14651858.CD007930.pub3. PMID 37185961

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Tivozanib | Standard Care
Started | 3 | 1
Completed | 3 | 1
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tivozanib | Standard Care | Total
Number analyzed (Participants) | 3 | 1 | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 1 | 3
  >=65 years | 1 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 4
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival (PFS) Comparison
Description: To compare progression-free survival of maintenance therapy with Tivozanib against standard of care in patients with ovarian, fallopian tube or primary peritoneal carcinoma who have achieved a complete response following therapy for platinum sensitive disease.
  Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1)
Time Frame: 2 Years
Population: Reporting the number of cycles each patient completed. Each cycle = 4 weeks.
Measure: Number; unit: Cycles
Arm/Group | Tivozanib | Standard Care
Number analyzed (Participants) | 3 | 1
Cycles
  Patient 1 | 6 | 0
  Patient 2 | 9 | 0
  Patient 3 | 2 | 0
  Patient 4 | 0 | 2

2. Secondary Outcome: Progression-Free Survival (PFS) Evaluation
Description: To evaluate progression-free survival with no maintenance therapy in patients who have achieved a complete response following therapy for platinum sensitive disease.
Time Frame: 2 Years
Population: Outcome measure not analyzed due to low accrual and subsequent termination of the study.
Arm/Group | Tivozanib | Standard Care
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Overall Survival (OS) Evaluation
Description: To evaluate the overall survival with and without maintenance therapy with Tivozanib in patients who have achieved a complete response following therapy for platinum sensitive disease.
Time Frame: 2 Years
Population: Outcome measure not analyzed due to low accrual and subsequent termination of the study.
Arm/Group | Tivozanib | Standard Care
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Toxicity Rate Comparison
Description: To compare rates of toxicity with and without maintenance therapy with Tivozanib.
Time Frame: 2 Years
Population: Outcome measure not analyzed due to low accrual and subsequent termination of the study.
Arm/Group | Tivozanib | Standard Care
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Quality of Life (QOL) Evaluation
Description: To evaluate the impact of treatment with Tivozanib versus placebo alone on the Quality of Life (QOL) through the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30) and the EORTC QLQ-Ovarian Cancer Module (EORTC QLQ-OV28) for functioning and symptoms.
Time Frame: 2 Years
Population: Outcome measure not analyzed due to low accrual and subsequent termination of the study.
Arm/Group | Tivozanib | Standard Care
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse event data was collected from the time of first treatment to 30 days after the last treatment.
Arm/Group | Tivozanib | Standard Care
Serious Adverse Events (participants affected / at risk) | 1/3 | 1/1
Other Adverse Events (participants affected / at risk) | 3/3 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tivozanib (N=3) | Standard Care (N=1)
Athralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tivozanib (N=3) | Standard Care (N=1)
Urinary tract pain (Renal and urinary disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Edema limbs (General disorders) | 1 (1) | 0 (0)
Athralgia (Musculoskeletal and connective tissue disorders) | 3 (8) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 2 (2) | 0 (0)
Skin infection (Infections and infestations) | 1 (1) | 0 (0)
Rash maculopapular (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 2 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 2 (2) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 3 (3) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (2) | 0 (0)
Dysgeusia (Nervous system disorders) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 1 (1)
Hypomagnesemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Memory impairment (Nervous system disorders) | 1 (1) | 0 (0)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0)
Chest pain - cardiac (Cardiac disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)
Vaginal pain (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hot flashes (Vascular disorders) | 1 (1) | 0 (0)
Urinary frequency (Renal and urinary disorders) | 1 (1) | 0 (0)
Bloating (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (2) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (3) | 0 (0)
Hypothyroidism (Endocrine disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (2) | 0 (0)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Terminated early due to low accrual.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less